CLINICAL TRIAL: NCT05211297
Title: Impact of Suspected Preterm Labour During Pregnancy on Cardiometabolic Profile and Neurodevelopment During Childhood: a Prospective Cohort Study Protocol.
Brief Title: Impact of Suspected Preterm Labour on Cardiometabolic Profile and Neurodevelopment
Acronym: SKs
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Cristina Paules, Principal Investigator, Instituto de Investigación Sanitaria Aragón
Other Study IDs: Superkids study
Record Dates: First submitted 2022-01-08; First posted 2022-01-27 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Preterm Labor
Keywords: pregnancy; preterm labor; neurodevelopment; cardiovascular; metabolic; prematurity
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed cohort:: Children whose mothers suffered a suspected preterm labour during pregnancy.
- Unexposed cohort: Children born at term (> 37 weeks) whose mothers did not suffer a suspected preterm labour during pregnancy.

SUMMARY:
Suspected preterm labour (SPL), define as the presence of regular and painful uterine contractions and cervical shortening, constitute a prenatal insult with potential long-term consequences. However, despite recent evidence demonstrating a suboptimal neurodevelopment at 2 years in this population, it remains under-recognized as a significant risk factor for neurodevelopmental disorders or other chronic diseases. The objective of this study is to assess the impact of suspected preterm labour during pregnancy on cardiometabolic profile and neurodevelopment during childhood (6-8 years).

Prospective cohort study including children whose mothers suffered a suspected preterm labor during pregnancy and paired controls. A neurodevelopment, cardiovascular and metabolic assessment at 6-8 years of age will be performed. A trained psychologist will carry out the neurodevelopment assessment. Body composition and physical fitness assessment will be performed by one trained pediatrician and nurse. Finally, cardiovascular assessment, including echocardiography and blood pressure, will be performed by two pediatric cardiologists. Data regarding perinatal and postnatal characteristics, diet, lifestyle and weekly screen time of the child will be obtained from clinical histories and direct interviews with the families. Primary outcome measures will include body mass index and adiposity, percentage of fat mass and total and regional lean mass, bone mineral content and density, cardio-respiratory resistance, isometric muscle strength, dynamic lower body strength, systolic and diastolic blood pressure, left ventricle (LV) systolic and diastolic function, general intelligence index, visuospatial working memory span, visual development test, visual acuity, index of emotional and behavioral problems.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Good understanding and sign of informed consent.

Exclusion Criteria:

* Multiple pregnancy
* Malformations
* Chromosomal diseases
* Prenatal infections

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Two cohorts of children at 6-8 years of age:
  A. Exposed cohort: children whose mothers suffered a suspected preterm labour during pregnancy. They are subdivided into:
  * Moderate-late preterm births (between 32 and 37 weeks of gestation)
  * "False suspected preterm labour" (full-term births (> 37 weeks) after suffering a suspected preterm labour) B. Unexposed cohort: children born at term (> 37 weeks) whose mothers did not suffer a suspected preterm labour during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Percentage of fat mass and total and regional lean mass | 6-8 years
Body mass index and adiposity | 6-8 years
Cardio-respiratory resistance | 6-8 years
  After fitting the safety harness, the test began when the participants were able to walk easily on the treadmill (Quasar Med 4.0, h/p/cosmos, Nußdorf, Germany). The protocol started with a speed of 2.4 km/h, increasing by 0.8 km/h every 2 min until the participants were unable to walk or reached a speed of 4.8 km/h. Then, the slope was increased by 4% every minute until exhaustion or up to a maximal slope of 24%. The respiratory gas exchange data were measured breath-by-breath using open-circuit spirometry (Oxycon Pro, Jaeger/Viasys Healthcare, Hoechberg, Germany). Maximal oxygen uptake (VO2max) values were averaged over consecutive 15 s periods.
Systolic and diastolic blood pressure | 6-8 years
Left ventricle (LV) systolic and diastolic function | 6-8 years
  End-diastolic and end-systolic diameter, septum and posterior wall thickness, heart rate, ejection fraction (by Teicholz and biplane Simpson methods), mitral annulus S´ wave velocity (tissue doppler), mitral annulus E and A waves velocity (pulse-wave doppler), E´ and A´ waves velocity (tissue doppler), TEI index (tissue doppler) and LV strain and strain rate at three apical views (speckle tracking).
General intelligence index | 6-8 years
Visual development test | 6-8 years
Global index of problems | 6-8 years
Index of emotional problems | 6-8 years
Index of behavioral problems | 6-8 years

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Paules, Principal Investigator — IISAragon . Clini Hospital Zaragoza.
Locations (1):
- Cristina Paules, Zaragoza, Aragon, Spain